CLINICAL TRIAL: NCT06878716
Title: Official Title : Silver Russell Syndrome, Parental Fertility and Assisted Reproductive Technology 600 caractères Maximum
Brief Title: Silver Russell Syndrome, Parental Fertility and Assisted Reproductive Technology
Acronym: SRS-AMP
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240670; IDRCB 2021-A02781-40 (Other: ANSM)
Record Dates: First submitted 2025-02-21; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Syndrome, Russell Silver
Keywords: Imprinting disorders; - Silver Russell syndrome; Infertility; Assisted Reproductive Technology; In vitro fertilization
MeSH Terms: conditions — Silver-Russell Syndrome; Imprinting Disorders; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Silver Russell Syndrome (SRS) is a rare imprinting disorder (about 1/16000). Parental imprinting is an epigenetic regulation phenomenon leading to the monoallelic expression of some genes. Its establishment takes place in the gametes and its maintenance is important at the early embryonic stage. Increase in the prevalence of conception by assisted reproductive technology (ART) has already been found in patients with imprinted disorder such as Angelman, Beckwith-Wiedemann or Prader Willi Syndromes, and more recently with SRS; ART is associated with an increase in the frequency of SRS. Several hypotheses are formulated to explain this increase. The first one is the involvement of the infertility etiology in the imprinting disorder genesis. The second one is the involvement of ART technics in the genesis of abnormal gamete imprinting during their manipulation or during imprinting maintenance at early embryonic stages.

Our main objective is to estimate ART conceptions prevalence in children followed for a SRS. The secondary objectives are to estimate infertility prevalence among parents of patients with SRS, to estimate factors frequency possibly responsible for the genesis of imprinting anomalies among parents of patients with SRS, to describe the infertility causes and to detail ART technics used (stimulation protocols, type of fertilization used, modality of embryonic culture and transfer, embryonic characteristics).

A transversal pilote study will be firstly conducted in parents of patients followed in Silver Russell Syndrome Reference Center (Pediatric Endocrine department, in Trousseau Hospital, Paris).

Data collection will be done by phone, after collecting the non-opposition of the parents, in order to complete a questionnaire concerning their fertility and conception mode of their child. If ART was used to conceive, a questionnaire concerning the details of the ART technics used will be sent to the doctor and:or the ART biologist, who performed the ART. The data will be anonymized and collected on a REDCap database.

DETAILED DESCRIPTION:
There is no planned follow-up, and the parents' participation is limited to the telephone interview.

The aim is to conduct / carry out a single-centre observational cross-sectional study, on the one hand by collecting data from the centre's patient files (molecular anomaly leading to the diagnosis of Silver Russell syndrome) and on the other hand by conducting a 30-minute telephone questionnaire to collect additional data. The first part of this questionnaire will be carried out with the parents of these patients in order to specify their age, height, weight, drug consumption and profession at the time of the start of pregnancy, as well as the time required for conception and recourse to ART.

In the event of recourse to ART, with the authorisation of the parent(s), a questionnaire will be sent to the clinical doctor and/or the biologist at the ART centre.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* parents from patients followed in the department " Unité Fonctionnelle Endocrinienne du Pr Netchine " for un Silver Russell syndrome

Exclusion Criteria:

* parent's objection
* patient under State Medical Aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children being followed for Silver-Russell syndrome at the Silver-Russell Syndrome Reference Centre at Trousseau Hospital in the Endocrine Functional Investigation Unit.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of SRS patients whose mode of conception was ART | Day 0, visit inclusion
  To estimate ART conceptions prevalence in children followed for a SRS

SECONDARY OUTCOMES:
Estimate infertility prevalence among parents of patients with SRS (defined as a delay to conception of more than 12 months) | Day 0, visit inclusion
  The time required for conception is defined by the time between stopping contraception and the start of pregnancy
Estimate frequency of maternal and paternal BMI at the time of conception | Day 0, visit inclusion
Estimate frequency of consumption of tobacco and alcohol at the time of conception | Day 0, visit inclusion
  At the time of conception maternal and paternal BMI, consumption of tobacco and alcohol and both parents' occupations
Estimate frequency of parents's profession at the time of conception | Day 0, visit inclusion
The etiology of infertility in detail | 3 years, end of the study
  Study infertility causes in detail this will be do through a questionnaire send to the fertility doctor who treated the parents.
Describe the ART techniques used from the point of view of ovarian stimulation but also oocyte, sperm and embryo manipulations | 3 years, end of the study
  Details of ART techniques used this will be do through a questionnaire send to the fertility doctor who treated the parents.

CONTACTS AND LOCATIONS:
Overall Officials: Irène Netchine, PUPH, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pediatric Endocrine department - Trousseau Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided